CLINICAL TRIAL: NCT00557648
Title: Early Interventions for Anxious Children
Brief Title: Evaluating the Effectiveness of Early Cognitive Behavioral Therapy With or Without Parental Involvement in Treating Anxious Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWA00000312-4; R21MH065369 (NIH)
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Children; Cognitive-Behavioral Therapy; School-Based Interventions
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): CBT for children only
  Interventions: Behavioral: Group CBT for children
- 2 (Experimental): CBT for children with parental involvement
  Interventions: Behavioral: Group CBT for children plus parent training
- 3 (No Intervention): No intervention control group: families free to seek treatment on their own

INTERVENTIONS:
Behavioral: Group CBT for children — CBT for children consists of 9 weekly group CBT sessions. All sessions occur in the school building during after-school hours.
  Arms: 1
Behavioral: Group CBT for children plus parent training — CBT involving children and parents consists of 9 weekly group CBT sessions for the children and 9 weekly concurrent group parent training sessions.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of school-based cognitive behavioral therapy with or without parental involvement in treating anxious children.

DETAILED DESCRIPTION:
Anxiety disorders are among the most common disorders in children. Although anxiety is a normal part of growing up, the worrying experienced by children with anxiety disorders can persist to the point that day-to-day functioning becomes difficult. Physical symptoms of anxiety disorders include a constant sense of worry or stress, headache, nausea, sweating, shaking, and inability to concentrate. Early identification of anxiety disorders is important to prevent progression of the disorder into a chronic issue. Cognitive behavioral therapy (CBT), which focuses on behavioral and thinking modifications, has been shown to be the most effective treatment for anxiety disorders. This study will evaluate the effectiveness of school-based CBT with or without parental involvement in treating anxious children who meet DSM-IV criteria or have features of separation anxiety disorder, generalized anxiety disorder, and social phobia.

Participants in this single blind study will be randomly assigned by school to one of three treatment groups: CBT for children only, CBT for children plus parent training, and no-treatment control. Each child and parent participant will first undergo an interview, lasting between 1 and 1.5 hours, about the child's symptoms. Additionally, parents will complete rating scales about their children's symptoms and their own symptoms. The participants receiving CBT will then attend 9 weekly group sessions held in the school buildings after school. In the parental involvement group, parents will attend 9 weekly group parent-training sessions held at the same time as the children's CBT group sessions. During the children's CBT sessions, participants will learn techniques to identify feelings of worry, relax, modify negative thoughts, break down difficult situations into smaller achievable steps, reward themselves for trying hard, and maintain treatment gains. For the parent training group, early sessions will focus on normalizing anxiety during childhood, learning about anxiety, and identifying when their children are feeling anxious. The middle sessions will teach parents the same anxiety management skills being taught to their children and ways to help their children to apply the steps at home. The latter sessions will instruct parents on ways to encourage their children's behaviors in anxiety-provoking situations. After completing the 9-week program, participants will attend 2 follow-up booster sessions at Months 1 and 3 post-treatment. Follow-up assessments will occur at Months 3 and 6 and at Years 1, 2, 3, and 4 post-treatment. The assessments will include repeat interviews and rating scales. At the end of the 6-month follow-up assessment, participants in the no-treatment control group will have the opportunity to participate in the CBT group treatments.

ELIGIBILITY:
Inclusion Criteria:

* Total Anxiety T-score of greater than 57 on Multidimensional Anxiety Scale for Children and/or teacher nomination as one of the most anxious children in the classroom
* Meets DSM-IV criteria for separation anxiety disorder, generalized anxiety disorder, and/or social phobia, or features (one or more, but not all criteria) of one of these disorders with an associated composite CSR of 2 to 6 on ADIS
* Both parent and child speak English fluently

Exclusion Criteria:

* Current diagnosis of the following on ADIS: obsessive-compulsive disorder, posttraumatic stress disorder, attention-deficit hyperactivity disorder, conduct disorder, schizophrenia, pervasive developmental disorder, major depression, or substance abuse
* Current suicidal or homicidal intent or plan
* Diagnosis of mental retardation (IQ less than 71) on the Kaufman Brief Intelligence Test (KBIT)
* Currently receiving psychotropic medication

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2002-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Composite Clinician Severity Rating (CSR) on the Anxiety Disorders Interview Schedule (ADIS) for DSM-IV for primary anxiety diagnosis | Measured at Month 6 and Years 1, 2, 3, and 4 post-treatment

SECONDARY OUTCOMES:
Multidimensional Anxiety Scale for Children, Scale for Child Anxiety Related Emotional Disorders, Clinical Global Impressions-Improvement Scale, Family Adaptability and Cohesion Evaluation Scale II, and Behavior Assessment System for Children | Measured at Months 3 and 6 and Years 1, 2, 3, and 4 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gail A. Bernstein, MD, Principal Investigator — Division of Child and Adolescent Psychiatry, University of Minnesota Medical School
Locations (1):
- Divisions of Child and Adolescent Psychiatry, University of Minnesota Medical School, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Bernstein GA, Layne AE, Egan EA, Tennison DM. School-based interventions for anxious children. J Am Acad Child Adolesc Psychiatry. 2005 Nov;44(11):1118-27. doi: 10.1097/01.chi.0000177323.40005.a1. PMID 16239860
- [Result] Bernstein GA, Layne AE, Egan EA, Nelson LP. Maternal phobic anxiety and child anxiety. J Anxiety Disord. 2005;19(6):658-72. doi: 10.1016/j.janxdis.2004.09.001. PMID 15927779
- [Result] Layne AE, Bernstein GA, March JS. Teacher awareness of anxiety symptoms in children. Child Psychiatry Hum Dev. 2006 Summer;36(4):383-92. doi: 10.1007/s10578-006-0009-6. PMID 16736381
- [Result] Victor AM, Bernat DH, Bernstein GA, Layne AE. Effects of parent and family characteristics on treatment outcome of anxious children. J Anxiety Disord. 2007;21(6):835-48. doi: 10.1016/j.janxdis.2006.11.005. Epub 2006 Dec 11. PMID 17161582
- [Result] Bernstein GA, Bernat DH, Davis AA, Layne AE. Symptom presentation and classroom functioning in a nonclinical sample of children with social phobia. Depress Anxiety. 2008;25(9):752-60. doi: 10.1002/da.20315. PMID 17557318
- [Result] Bernstein GA, Bernat DH, Victor AM, Layne AE. School-based interventions for anxious children: 3-, 6-, and 12-month follow-ups. J Am Acad Child Adolesc Psychiatry. 2008 Sep;47(9):1039-47. doi: 10.1097/CHI.ob013e31817eecco. PMID 18665000
- [Result] Layne AE, Bernat DH, Victor AM, Bernstein GA. Generalized anxiety disorder in a nonclinical sample of children: symptom presentation and predictors of impairment. J Anxiety Disord. 2009 Mar;23(2):283-9. doi: 10.1016/j.janxdis.2008.08.003. Epub 2008 Aug 12. PMID 18815006